CLINICAL TRIAL: NCT04225858
Title: Avoiding Sentinel Lymph Node Biopsy In Select Clinical Node Negative Breast Cancer Patients After Neoadjuvant Systemic Therapy: the ASICS Trial
Brief Title: Avoiding Sentinel Lymph Node Biopsy in Breast Cancer Patients After Neoadjuvant Chemotherapy
Acronym: ASICS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N19ASC
Record Dates: First submitted 2019-12-04; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; HER2-positive Breast Cancer; Sentinel Lymph Node
Keywords: Neoadjuvant Chemotherapy; Sentinel lymph node biopsy; Breast cancer; Complete response
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Intervention Model Description: Prospective non-inferiority cohort, single-arm registration trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omission of sentinel lymph node biopsy (Experimental): No surgical axillary staging (i.e. sentinel lymph node biopsy) will be performed.
  Interventions: Procedure: Omission of sentinel lymph node biopsy

INTERVENTIONS:
Procedure: Omission of sentinel lymph node biopsy — No sentinel lymph node biopsy will be performed in clinically node-negative triple-negative or HER2-positive breast cancer patients with a radiologic complete response on MRI. Participants will be asked to complete quality of life questionnaires at baseline (prior to surgery), 6 months, 1, 3 and 5 years follow-up. A control group consisting of 100 clinically node-negative patients receiving standard treatment will be used to compare QoL scores. This group consists of patients that do not wish to participate in the experimental group (i.e., no sentinel node lymph node biopsy) or patients that are not eligible.
  Other Names: Quality of life assessment

SUMMARY:
This study evaluates whether SLNB can safely be omitted in breast cancer patients with HER2+ or TN tumors who achieve a radiological complete response on MRI after neoadjuvant systemic therapy

DETAILED DESCRIPTION:
Axillary staging in clinically node negative (cN0) breast cancer patients with neoadjuvant systemic therapy (NST; i.e. chemo- and immunotherapy), is preferably performed with sentinel lymph node biopsy (SLNB) after NST. The probability of a tumor-positive SLNB post-NST is low. cN0 patients with Human Epidermal growth factor Receptor 2- positive (HER2+) or triple negative (TN) breast cancer who achieve radiologic complete response (rCR) of the breast on MRI, have the lowest probability of a tumor-positive SLNB post-NST (<3%). Omitting removal of axillary lymph nodes in clinically node negative patients does not increase the rate of distant metastases nor breast cancer mortality. Performing SLNB can cause short- and long-term morbidity, reducing quality of life. The additional value of performing SLNB in patients with a very low risk of tumor-positive axillary lymph nodes should be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged ≥ 18 years
* Invasive HER2+ (HR+/-) or TN breast cancer
* Primary tumor (T), clinical stage T1-3
* Neoadjuvant systemic therapy (NST), at least 3 cycles
* Tumor stage assessed with breast MRI before start NST
* Clinically node-negative before start NST (no suspect ALNs on ultrasound and FGD-PET/CT, or negative cyto-/histopathology in case of suspect nodes)
* MRI after or during NST shows radiologic complete response
* Written and signed informed consent

Exclusion Criteria:

* Primary tumor (T) clinical stage T4
* Patients without ultrasound or FDG-PET/CT pre-NST
* History of breast cancer ipsilateral breast
* Synchronous contralateral breast cancer
* Synchronous M1 disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Axillary recurrence | at 5 years
  To show that sentinel lymph node biopsy after neoadjuvant systemic therapy can be omitted in clinically node-negative HER2+ or TN breast cancer patients who achieve radiological complete response on MRI without compromising the 5 - year axillary recurrence rate (i.e, < 6% axillary recurrences within 5 years).

SECONDARY OUTCOMES:
Breast cancer specific quality of life | at 5 years
  To compare study participants in whom sentinel lymph node biopsy is omitted to patients with sentinel lymph node biopsy on breast cancer related quality of life, especially axillary morbidity score. This is measured with the EORTC-BR23 scale. The arm morbidity score consists of 3 items, points ranging from 1 - 4 per item. A higher score indicates more morbidity.
Level of cancer worry | at 5 years
  To compare study participants in whom sentinel lymph node biopsy is omitted to patients with sentinel lymph node biopsy on level of cancer worry, using the cancer worry scale (CWS). The CWS consists of 8 items, with 1-4 points per item and a maximum score of 32 points. Higher scores indicate more frequent cancer worry.
Recurrence-free survival | at 5 years
  To assess 5-year recurrence-free survival in clinically node-negative HER2+ or TN patients with radiologic complete response on MRI in whom sentinel lymph node biopsy is omitted.
Overall survival | at 5 years
  To assess 5-year overall survival in clinically node-negative HER2+ or TN patients with radiologic complete response on MRI in whom sentinel lymph node biopsy is omitted.
Disease-specific survival | at 5 years
  To assess 5-year disease specific survival in clinically node-negative HER2+ or TN patients with radiologic complete response on MRI in whom sentinel lymph node biopsy is omitted.

OTHER OUTCOMES:
Axillary recurrence rate by pathological response | at 5 years
  To assess 5-year axillary recurrence-free survival in patients with and without a pathological complete response
Recurrence rate by pathological response | at 5 years
  To assess 5-year recurrence-free survival in patients with and without a pathological complete response
Survival by pathological response | at 5 years
  To assess 5-year survival in patients with and without a pathological complete response

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Jeanne T.F.D. Vrancken Peeters, MD, PhD, Principal Investigator — Antoni van Leeuwenhoek